CLINICAL TRIAL: NCT03516708
Title: Phase I/II Study of Epacadostat (INCB024360) Added to Preoperative Chemoradiation in Patients With Locally Advanced Rectal Cancer
Brief Title: Epacadostat (INCB024360) Added to Preoperative Chemoradiation in Patients With Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202305133 (201902040); 1R01CA278197 (NIH)
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer
Keywords: Immunotherapy; Kynurenine; Colon; Indoleamine 2,3 dioxygenase; IDO1
MeSH Terms: conditions — Rectal Neoplasms | interventions — epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation Cohort (Phase I): Epacadostat + SCRT + Chemotherapy + Surgery (Experimental): * Epacadostat at the designated dose level starting on the 1st day of radiation therapy and continuing throughout chemotherapy until the day of surgery.
  * Standard of care preoperative therapy will consist of a total of approximately 20-24 weeks of short-course pelvic radiation and chemotherapy:
    * Cycle 0 Days 1-7(Week 1): Short-course pelvic radiation therapy (SCRT), 5 fractions over 1 week
    * Cycle 0 Days 8-21 or 8-28 (Weeks 2-4): Treatment break for 2 to 3 weeks; for patients enrolled at Washington University and Dana Farber only, tumor biopsy will be obtained between the end of RT and prior to chemotherapy (target Days 14-28)
    * Cycles 1-6: (6) 21-day cycles of CAPOX for a total of 18 weeks. CAPOX is typically capecitabine at 1000 mg/m^2 PO BID (days 1-14 of each cycle) and oxaliplatin 130 mg/m^2 IV Q3W.
    * Surgery will follow approximately 4 to 6 weeks after completion of CAPOX
  Interventions: Drug: Epacadostat; Radiation: Short-course radiation therapy; Drug: CAPOX chemotherapy
- Phase II Treatment Cohort: Epacadostat + SCRT + Chemotherapy + Surgery (Experimental): * Epacadostat 400 mg BID 1st day of radiation therapy and continuing for ~28 days, until biopsy (with the exception of patients enrolling to dose expansion and starting on epacadostat with neoadjuvant chemotherapy prior to approval of post-sIRB A2)
  * Preoperative therapy approximately 20-24 weeks of chemoradiation:
    * Week 1: SCRT, typically 5 Gy x 5 fractions over 1 week, with epacadostat 400 mg BID starting on D1 of SCRT
    * Weeks 2-4: Epacadostat monotherapy 400 mg BID & continued for a minimum of 21 days, until the day prior to chemotherapy
    * For patients enrolled at Washington University and Dana Farber Cancer Institute ONLY, tumor biopsy between the end of RT and prior to initiation of chemotherapy. Tumor biopsy target of between Days 15-28
    * Weeks 3-6: 4-5 weeks after completion of SCRT & after completion of approximately 21-35 days of epacadostat, SOC neoadjuvant chemotherapy of CAPOX or FOLFOX will be initiated
    * Surgery will occur approximately 4-6 weeks after chemotherapy
  Interventions: Drug: Epacadostat; Radiation: Short-course radiation therapy; Drug: CAPOX chemotherapy; Drug: FOLFOX chemotherapy
- Phase II Biomarker Cohort: SCRT + Chemotherapy + Surgery (Active Comparator): Washington University and Dana Farber only: Patients enrolled to this cohort will not receive epacadostat. Patients will undergo standard of care preoperative therapy consisting of approximately 20 to 24 weeks of chemoradiation. All treatment will be administered in this cohort as per institutional standard. The expected schedule for these patients will consist of 1 week of short-course pelvic radiation therapy, followed by a treatment break, followed by neoadjuvant chemotherapy. Approximately 4 to 6 weeks after completion of neoadjuvant chemotherapy, patients may undergo surgery. Tumor biopsy may occur at screening and after completion of RT, prior to starting neoadjuvant chemotherapy.
  Interventions: Radiation: Short-course radiation therapy; Drug: CAPOX chemotherapy; Drug: FOLFOX chemotherapy

INTERVENTIONS:
Drug: Epacadostat — Drug provided.
  Other Names: INCB024360
  Arms: Dose Escalation Cohort (Phase I): Epacadostat + SCRT + Chemotherapy + Surgery; Phase II Treatment Cohort: Epacadostat + SCRT + Chemotherapy + Surgery
Radiation: Short-course radiation therapy — Short-course pelvic radiation therapy, 5 Gy x 5 fractions over 1 week
  Other Names: SCRT
Drug: CAPOX chemotherapy — Standard of care
Drug: FOLFOX chemotherapy — Standard of care
  Arms: Phase II Biomarker Cohort: SCRT + Chemotherapy + Surgery; Phase II Treatment Cohort: Epacadostat + SCRT + Chemotherapy + Surgery

SUMMARY:
The purpose of this research study is to evaluate epacadostat when given with routine radiation therapy and chemotherapy (capecitabine and oxaliplatin) to treat rectal cancer before routine surgery is performed to remove the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pathologically-confirmed locally advanced rectal cancer (defined by 8th edition AJCC stage 2 or 3, or stage 1 not eligible for sphincter-sparing surgery) with plans to proceed with total neoadjuvant short course radiation as part of their neoadjuvant therapy as confirmed by treating physician
* At least 18 years of age.
* ECOG performance status 0, 1, or 2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin > 9 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Serum creatinine < 1.5 x IULN OR measured or calculated creatinine clearance ≥ 50 mL/min/1.73 m2
* Applicable to subjects enrolled at Washington University and Dana Farber Cancer Institute only: Willing to undergo study-related biopsies subject to accessibility of tumor, appropriateness of biopsy (not contraindicated), and continued subject consent. If biopsy is not safe and feasible per treating physician, then patient may still enroll with permission of sponsor-investigator.
* Women of childbearing potential and men must agree to contraceptive methods as described in protocol prior to study entry, for the duration of study participation, and for 120 days after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Received prior anti-cancer therapy for rectal cancer.
* Prior treatment with agents targeting IDO pathway (including indoximod)
* Previous radiotherapy in the pelvic region or previous rectal surgery (e.g. TEM) or any investigational treatment for rectal cancer within the past month.
* Known or suspected presence of another malignancy that could be mistaken for the malignancy under study during disease assessments.
* Currently receiving any other investigational agents.
* Extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumor downsizing is seen.
* Presence of metastatic disease or recurrent rectal tumor.
* Diagnosis of Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease, or active ulcerative colitis.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to epacadostat, pembrolizumab, 5-FU, oxaliplatin, or other agents used in the study.
* Has an active infection requiring systemic therapy.
* Warfarin (Coumadin): patients currently on warfarin are excluded. Patients who go off warfarin and have INR within normal limits have no washout period.
* Any history of serotonin syndrome (SS) after receiving serotonergic drugs. This syndrome has been most closely associated with the use of MAOIs, meriperidine, linezolid, or methylene blue; all of these agents are prohibited during the study
* Uncontrolled intercurrent illness including, but not limited to active tuberculosis infection, pneumonitis requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Has an active or inactive autoimmune disease or syndrome (i.e. rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) that has required systemic treatment in the past 2 years or is receiving systemic therapy for an autoimmune or inflammatory disease (i.e. with use of modifying agents, corticosteroids, or immunosuppressive drugs). Exceptions include subjects with vitiligo or resolved childhood asthma/atopy, hypothyroidism stable on hormone replacement, controlled asthma, Type I diabetes, Graves' disease, or Hashimoto's disease.
* An abnormal screening ECG that, in the investigator's opinion, is clinically meaningful.
* Presence of a gastrointestinal condition that may affect drug absorption.
* Receipt of live attenuated vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of planned start of study therapy.
* Known active hepatitis B (e.g. HBsAg reactive or HBV DNA detected) or hepatitis C (e.g. HCV RNA [qualitative] is detected) infection. Testing at screening is required (Serology testing with HBsAg, HBsAb, and HCV Ab are required; HBV DNA or HCV RNA are only required in the setting of serology tests compatible with possible active infection.).
* Known microsatellite instability- high (MSI-H) or mismatch repair deficient rectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2030-08-12 (Estimated)

PRIMARY OUTCOMES:
Phase I only: Recommended phase II dose (RP2D) of epacadostat with standard of care radiation and chemotherapy in preoperative treatment of locally advanced rectal cancer | Completion of the first 2 cycles of treatment for all patients (estimated to be 86 months)
  The recommended phase 2 dose (RP2D) is defined as the dose level immediately below the maximally administered dose at which 0 or 1 of a cohort of 3 to 6 patients experienced a dose-limiting toxicity (DLT) during first 2 cycles.
Phase II Treatment Cohort only: Neoadjuvant Rectal (NAR) Score | At the time of surgery (approximately week 28)
  Neoadjuvant Rectal Score (NAR Score) is calculated by following formula: NAR = ([5pN
  - 3(cT - pT) + 12]2)/9.61 (with higher scores representing poorer prognosis), where cT=clinical tumor stage, pT=pathologic tumor stage, and pN=pathologic nodal stage.

SECONDARY OUTCOMES:
Phase I and Phase II Treatment Cohort only: Safety and toxicity profile of the combination as measured by adverse events experienced | Through 4 weeks after completion of treatment (approximately 28 weeks)
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Phase I only: Neoadjuvant Rectal (NAR) Score | At the time of surgery (approximately week 28)
  Neoadjuvant Rectal Score (NAR Score) is calculated by following formula: NAR = ([5pN
  - 3(cT - pT) + 12]2)/9.61 (with higher scores representing poorer prognosis), where cT=clinical tumor stage, pT=pathologic tumor stage, and pN=pathologic nodal stage.
Phase I and Phase II Treatment Cohort only: Pathological complete response rate (pCR) | At the time of surgery (approximately week 25)
  Pathologic complete response (pCR) is defined as no histology evidence of invasive tumor cells in the surgical specimen.
Phase I and Phase II Treatment Cohort only: Progression-free survival (PFS) | Through completion of follow-up (estimated to be 3 years and 32 weeks)
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. For those who are alive and do not experience progression, they are censored at the time of loss to follow-up.
Phase I and Phase II Treatment Cohort only: Complete clinical response rate (cCR) | At the time of preoperative assessment (approximately week 28)
  Clinical complete response (cCR) is defined as no clinical evidence of tumor as assessed by radiographic, endoscopic, and physical examinations after completion of planned protocol therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Moh'd Khusman, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of California Irvine - Chao Family Comprehensive Cancer Center, Orange, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu